CLINICAL TRIAL: NCT06373978
Title: A Randomized Controlled Trial: Alternative Post Procedural Analgesia With NSAIDs vs Opioids in Percutaneous Needle Tenotomy of Elbow
Brief Title: NonNarcotic Pain Control in Percutaneous Needle Tenotomy of Elbow
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Michael Dakkak, Study PI, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 24-307
Record Dates: First submitted 2024-04-01; First posted 2024-04-18 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Elbow Pain; Chronic Pain
Keywords: TenJet; Elbow
MeSH Terms: conditions — Chronic Pain | interventions — Diclofenac; Tramadol; Acetaminophen

STUDY DESIGN:
Intervention Model Description: This study is a double-blind, randomized controlled trial comparing the effectiveness of oral acetaminophen, diclofenac, and tramadol in reducing the consumption of narcotic doses (primary outcome) and minimizing patients' exposure to narcotics (secondary outcome) following an ultrasound-guided percutaneous needle tenotomy procedure on the lateral elbow.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Diclofenac (Active Comparator): 50mg
  Interventions: Drug: Diclofenac; Other: Acetaminophen
- Tramadol (Active Comparator): 50mg
  Interventions: Drug: Tramadol; Other: Acetaminophen
- Acetaminophen (Sham Comparator): 1000mg
  Interventions: Other: Acetaminophen

INTERVENTIONS:
Drug: Diclofenac — 50mg every 8hours as needed for pain
  Arms: Diclofenac
Drug: Tramadol — 50mg every 8hours as needed for pain
  Arms: Tramadol
Other: Acetaminophen — 1000mg every 8hours as needed for pain

SUMMARY:
This study is a double-blind, randomized controlled trial comparing the effectiveness of oral acetaminophen, diclofenac, and tramadol in reducing the consumption of narcotic doses (primary outcome) and minimizing patients' exposure to narcotics (secondary outcome) following an ultrasound-guided percutaneous needle tenotomy procedure on the lateral elbow.

DETAILED DESCRIPTION:
Tramadol is currently the standard post-procedure medication. Acetaminophen will be prescribed (1000 mg) and should be taken every 8 hours if pain is present. Tylenol should be the first taken for pain. If pain persist, the study kit containing the blinded, pain-controlled capsules will be taken second. Both diclofenac potassium (50mg) and tramadol (50mg) will be provided in identical-looking capsules and randomly assigned to patients in sealed packets by a physician, ensuring the double-blind nature of the study and be instructed to use every 8 hours as needed for pain If pain is still not adequately controlled an hour after taking the blinded study pack, a rescue medication, consisting of tramadol 50mg capsules, will also be supplied to the NSAID group in sealed packets while rescue medication of oral diclofenac will be provided to the opioid group. These medications will be administered immediately after the tenotomy procedure to all participants. The primary endpoint of the study will be the total count of tramadol doses taken by each group at the 10 day (± 4 days) postoperative follow-up. Pill counts from sealed packages and the use of rescue narcotics will be verified during the in-person visit at 10 days (± 4 days) .

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Male or female, aged 18-65 years
* Percutaneous Needle Tenotomy of Lateral Elbow Procedure
* Ability to take oral medication and willingness to participate in a 2-week follow-up pill counts
* Musculoskeletal ultrasound or MRI with diagnosis of tendinosis of the common extensor tendon of the elbow

Exclusion Criteria:

* • Any full thickness common extensor tendon tear of the elbow

  * Prior history of elbow surgery
  * Symptomatic cervical radiculopathy
  * Concurrent symptoms of the medial elbow
  * Treatment with another investigational drug or other intervention concurrently or previously that would interfere with postoperative pain control
  * Psychiatric illness that impedes evaluation of pain and/or narcotics use
  * No history of inflammatory arthritis, diabetes, chronic regional pain syndrome, connective tissue disease, fibromyalgia or autoimmune disease
  * No contraindications to NSAIDs or Opioids

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2024-08-12 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Number of pills taken | 10 days
  The number of total Tramadol pills taken per patient between the control (Tramadol + Diclofenac rescue) vs experimental (Diclofenac + Tramadol rescue) groups at two weeks.

SECONDARY OUTCOMES:
Non narcotic use | 10 days
  The percentage of patients randomized to Diclofenac that do not use any narcotic (Tramadol) rescue medication

CONTACTS AND LOCATIONS:
Overall Officials: Michael Dakkak, DO, Principal Investigator — Cleveland Clinic Florida
Locations (2):
- United States (2):
  - The Cleveland Clinic Florida, Coral Springs, Florida
  - The Cleveland Clinic Ohio, Avon, Ohio

IPD SHARING:
Plan to Share IPD: No